CLINICAL TRIAL: NCT06998888
Title: Determining the Effectiveness of Remote Monitoring of Cancer Patients Undergoing Outpatient Oral Cancer Treatment Using Caaring® Software
Brief Title: Determining the Effectiveness of Remote Monitoring of Cancer Patients With Oral Cancer Treatment Using Caaring® Software
Acronym: ONCOCAARING
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Persei Vivarium (Other)
Collaborators: Effice Servicios Para la Investigacion S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ONCOCAARING
Record Dates: First submitted 2025-05-21; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Cancer
Keywords: Caaring; Digital Care; Cancer; Remote patient monitoring; Online telemonitoring; DTx
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online telemonitoring group (G_CAARING) (Active Comparator): The monitoring and control of these patients will be carried out remotely through the Caaring® platform. Patients will connect to an APP on a mobile phone. They will have to complete the data and questionnaires related to the study variables.
  Interventions: Device: software Caaring (remote monitoring app)
- Control Group (G_Control) (No Intervention): The data of these patients are collected prospectively from their routine medical visits for 12 weeks after inclusion

INTERVENTIONS:
Device: software Caaring (remote monitoring app) — Caaring is an electronic data collection notebook that allows patients to confidentially fill out data/ questionnaires on their mobile phone and report them through an application that will be installed on the patient's mobile phone. Besides, This group (G_CAARING) will receive educational and prevention recommendations relative to cancer.
  Arms: Online telemonitoring group (G_CAARING)

SUMMARY:
The goal of this clinical trial investigation with device is to determinate the efficacy of the remote monitoring in cancer patients with a software called Caaring® a través del cumplimento terapéutico y de dosis.

The main question it aims to answer is if the development of a self-management platform (Caaring®) empowers cancer patients throughout their illness, reducing the number of in-person and telephone visits assisted by specialized medical and nursing staff. For this, researchers will compare the assessments between the two groups.

This is a randomized study with two arms. Online telemonitoring group: The follow-up of these patients will be carried out prospectively remotely through the Caaring® platform. And Prospective Control group: The data of these patients are collected prospectively for their routine medical visits for 12 weeks after their inclusion.

Caaring group patients must have sufficient technological skills to use a smartphone.

DETAILED DESCRIPTION:
This is a longitudinal, comparative non-inferiority, multicenter, with 2 arms Medical Device Clinical Trial.

The protocol and informed consent documents have been reviewed and approved by the hospital human subjects reviewboard and the study will be performed in accordance with the Declaration of Helsinki

ELIGIBILITY:
Inclusion Criteria:

* Patients who provide informed consent.
* Age ≥18 years.
* Oncology patients undergoing active outpatient oral therapy with: capecitabine, cyclin inhibitors, hormonal therapies, TKI inhibitors, monotherapy with or without intravenous therapy.
* Oncology patients undergoing active outpatient oral oncology treatment expected within 12 weeks of inclusion.
* Patients who must demonstrate sufficient technological skills to operate a smartphone through the "technological skills questionnaire."
* Patients who do not meet the exclusion criteria.

Exclusion Criteria:

* Patients with cognitive or sensory difficulties or insufficient command of Spanish language that, in the opinion of the healthcare professional conducting the recruitment, makes it difficult to understand the questions posed in the surveys, scales, or instruments used in the study, provided they do not have a legal representative capable of participating in the study.
* Patients for whom it is anticipated that follow-up will not be possible due to a change of residence.
* Patients who are participating in any other clinical trial or experimental study at the time of recruitment. Participation in observational studies will not be an exclusion criteria.
* Patients whose primary diagnosis is a mental illness or another poorly controlled medical condition.
* Terminally ill patients and/or those receiving palliative care according to the criteria of SECPAL (Spanish Society of Palliative Care).
* Institutionalized patients.
* Patients who, according to the recruiting professional's assessment, are not considered eligible for inclusion because they are undergoing specific follow-up care in other units (hemodialysis, transplants, etc.) requiring mandatory hospital visits less frequently than once every two months.
* Patients who do not demonstrate sufficient technological skills to use a smartphone through the "technological skills questionnaire."

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of adherence to treatment prescribed for cancer | 12 weeks
  The Percentage of adherence to treatment prescribed for cancer will be calculed: Units minus unused units, multiplied by 100

SECONDARY OUTCOMES:
Percentage of patients with al least 80% of data completed | Week 12
  Percentage of patients with al least 80% of data completed in the application.
Percentage of patients with 100% of data completed | Week 12
  Percentage of patients with 100% of data completed in the application
Changes in the use of health resources | Day 0 and Monthly up to 12 weeks
  Change in patient´s use of health resources scores al basal monthly and at the end of the study compared to baseline: Number of visits to specialist (e.g. oncology, primary care etc), number of emergency room vistis or number of new hospitalizations.
Patient satisfaction with the software Caaring | Week 12
  The patient satisfaction will be measured through a specific satisfaction questionnaire created for this purpose. Values: 3-15, a higher score refletcs greater satisfaction with software care.

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital Universitario HM Monteprincipe, Boadilla del Monte, Madrid
  - Hospital Universitario HM Sanchinarro, Hortaleza, Madrid
  - Hospital Universitario HM Puerta del Sur, Móstoles, Madrid

IPD SHARING:
Plan to Share IPD: No